CLINICAL TRIAL: NCT05500911
Title: Evaluation of a Bioactive Surface in Posterior Maxillary Sites: Controlled Clinical Trial
Brief Title: Bioactive Surfaces vs. Conventional Surfaces in Implants Placed in Atrophic Maxilla With Simultaneous Sinus Lift
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo (Other)
Responsible Party: Principal Investigator, Luigi Canullo, Principal investigator, Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT2
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Edentulous; Alveolar Process, Atrophy; Edentulous Alveolar Ridge Atrophy
Keywords: dental implant; implant surface; sinus lift; sinus floor elevation
MeSH Terms: conditions — Mouth, Edentulous; Atrophy

STUDY DESIGN:
Intervention Model Description: After the sinus lift procedure (performed with OSSIX® BONE on all study subjects), control group will be treated with a traditional implant surface (MultiNeO CS), test group will be treated with a bioactive surfaced implant (NINA MultiNeO NH)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NINA- MultiNeO NH (Active Comparator): After the sinus lift procedure (performed with OSSIX® BONE on all study subjects) treatment group will be treated with a bioactive surfaced implant (NINA MultiNeO NH)
  Interventions: Procedure: sinus lift; Procedure: implant placement
- MultiNeO CS (Active Comparator): After the sinus lift procedure (performed with OSSIX® BONE on all study subjects) control group will be treated with a traditional implant surface (MultiNeO CS)
  Interventions: Procedure: sinus lift; Procedure: implant placement

INTERVENTIONS:
Procedure: sinus lift — when residual bone height is >4 mm sinus lift through crestal approach procedure will be performed and after sinus flor elevation, OSSIX® Bone will be placed in the sinus cavity.
  Other Names: sinus floor elevation
Procedure: implant placement — Implant will be placed in edentulous area

SUMMARY:
In this controlled clinical study, a maxillary sinus lift (crestal approach) with OSSIX® Bone will be performed, and then implants MultiNeO CS (control group) and NINA MultiNeO NH (test group) will be inserted in edentulous posterior maxillae of study subjects. .+the clinical and radiographic results of the rehabilitation of posterior edentulous maxillary areas, obtained with traditional surface implants (MultiNeO CS, control group), are compared with those obtained with bioactive surface implants (NINA - MultiNeO NH, test group ).

DETAILED DESCRIPTION:
In this post- market controlled clinical study, the tested CE-marked dental implants are MultiNeO CS 1930 and NINA MultiNeO NH 9330, both manufactured by Alpha-Bio Tec. NeO or MultiNeO is defined as a system since it includes three types of connections: a conical narrow connection (CHC), a conical standard conical connection (CS) and an Internal Hex connection (IH). The fixture has a straight coronal part, a slightly tapered body, and a conical apical part. We will use MultiNeO CS to treat control group. One of the MultiNeO CS biggest clinical advantages since it is as good at bone type 4 as it is at bone type 1, 2 or 3.

MultiNeO CS has an implant surface with a sub-micron scale roughness created by Aluminum oxide blasting and double acid etching.

NINA MultiNeO NH is used for tret group, it has got an innovative bioactive surface.

NINA MultiNeO NH surface is a combination of the abovementioned roughening process and the creation of titanium oxide nano structure. Its hydrophilic part is created by resorbable salt thus maintaining its hydrophilicity Patient requiring sinus floor elevation with native bone crest height > 4 mm will be enrolled.Although a variety of implant surface are available for implant supported rehabilitation, the first hypothesis is that NINA MultiNeO NH Alpha-Bio Tec will be present faster osteointegration time compared to MultiNeO CS when adopted to rehabilitate of missing teeth in case of critical areas such as in the posterior mandible with critical bone defects. The second hypothesis is that NINA MultiNeO NH will promote a better apical bone regeneration in patients treated with sinus lift compared to MultiNeO CS due to its bioactive surface.

ELIGIBILITY:
Inclusion Criteria:

* edentulous posterior maxillae
* residual bone height > 4mm
* healthy periodontal conditions

Exclusion Criteria:

* smokers over 5 cigarettes/day
* Pregnancy (confirmed by verbal inquiry)
* Chronic systemic pathologies and neoplastic of the Oro-Facial District
* bisphosphonates intake
* Any sites where an implant already failed sites
* Untreated Periodontitis
* Sites with acute infections
* Chronic inflammatory diseases of the oral cavity
* Autoimmune diseases (cortisone intake)
* Allergy declared to one or more medicaments to be used during treatment
* Alcoholics patients and/or drug addicts
* collagen hypersensitivity.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Marginal bone change | 6 months after implant placement
  radiographic evaluation of the marginal bone level around the implant using a periapical x ray. marginal bone loss is in millimeters and indicates how many millimeters of bone has been lost
Marginal bone change | 12 months after implant placement
  radiographic evaluation of the marginal bone level around the implant using a periapical x ray. marginal bone loss is in millimeters and indicates how many millimeters of bone has been lost
Implant stability | immediately after implant placement
  check implant stability using resonant frequency analysis (RFA) Resonance frequency analysis (RFA) provides objective measurements of implant stability in a non-invasive way on the bone-implant interface. The results of the resonance frequency analysis are transformed into implant stability quotient (ISQ) values. ISQ, implant stability quotient, depends on the transducer used and is recorded as a number between 1 and 100, 100 representing the highest degree of stability. Transducers are designed for specific implant types and calibrated by the manufacturer.
Implant stability | 2 months after implant placement
  Resonance frequency analysis (RFA) provides objective measurements of implant stability in a non-invasive way on the bone-implant interface. The results of the resonance frequency analysis are transformed into implant stability quotient (ISQ) values. ISQ, implant stability quotient, depends on the transducer used and is recorded as a number between 1 and 100, 100 representing the highest degree of stability. Transducers are designed for specific implant types and calibrated by the manufacturer.
Implant stability | 4 months after implant placement
  Resonance frequency analysis (RFA) provides objective measurements of implant stability in a non-invasive way on the bone-implant interface. The results of the resonance frequency analysis are transformed into implant stability quotient (ISQ) values. ISQ, implant stability quotient, depends on the transducer used and is recorded as a number between 1 and 100, 100 representing the highest degree of stability. Transducers are designed for specific implant types and calibrated by the manufacturer.
insertion torque curve | During implant placement (T0 baseline
  The Insertion torque data were recorded and exported as a curve The torque curve records the amount of energy that was needed for arrive at the positioning of the implant.
  unit of measurement of torque is Newton centimeter (Ncm)

SECONDARY OUTCOMES:
Apical Bone regeneration | 6 months after implant placement
  Apical bone regeneration is calculated by the difference in volume between CBCT at baseline and 6 months follow-up
Evaluation the effects of bioactive implant surface (NINA- MultiNeO NH) in Apical Bone regeneration performed under the schneiderian membrane lining the maxillary sinus. Apical Bone regeneration defines the osseoinductive potential of a surface. | 12 months after implant placement
  Apical bone regeneration is calculated by the difference in volume between CBCT at baseline and 6 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Studio Odont.Associato Dr.P.Cicchese E L.Canullo, Rome, Italy/Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gittens RA, Scheideler L, Rupp F, Hyzy SL, Geis-Gerstorfer J, Schwartz Z, Boyan BD. A review on the wettability of dental implant surfaces II: Biological and clinical aspects. Acta Biomater. 2014 Jul;10(7):2907-18. doi: 10.1016/j.actbio.2014.03.032. Epub 2014 Apr 5. PMID 24709541
- [Background] Han J, Lulic M, Lang NP. Factors influencing resonance frequency analysis assessed by Osstell mentor during implant tissue integration: II. Implant surface modifications and implant diameter. Clin Oral Implants Res. 2010 Jun;21(6):605-11. doi: 10.1111/j.1600-0501.2009.01909.x. PMID 20666787
- [Background] Oates TW, Valderrama P, Bischof M, Nedir R, Jones A, Simpson J, Toutenburg H, Cochran DL. Enhanced implant stability with a chemically modified SLA surface: a randomized pilot study. Int J Oral Maxillofac Implants. 2007 Sep-Oct;22(5):755-60. PMID 17974109
- [Background] Pjetursson BE, Lang NP. Sinus floor elevation utilizing the transalveolar approach. Periodontol 2000. 2014 Oct;66(1):59-71. doi: 10.1111/prd.12043. PMID 25123761
- [Background] Stacchi C, Lombardi T, Ottonelli R, Berton F, Perinetti G, Traini T. New bone formation after transcrestal sinus floor elevation was influenced by sinus cavity dimensions: A prospective histologic and histomorphometric study. Clin Oral Implants Res. 2018 May;29(5):465-479. doi: 10.1111/clr.13144. Epub 2018 Mar 23. PMID 29569763